CLINICAL TRIAL: NCT00777868
Title: A Dose-Ranging Study Evaluating the Safety and Efficacy of IDP-108 in Patients With Onychomycosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dow Pharmaceutical Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DPSI-IDP-108-P2-01
Record Dates: First submitted 2008-10-20; First posted 2008-10-22 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2012-06

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: Low Strength IDP-108
- 2 (Experimental)
  Interventions: Drug: High Strength IDP-108
- 3 (Experimental)
  Interventions: Drug: High Strength IDP-108 under occlusion
- 4 (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Low Strength IDP-108 — Topical application once a day for 9 months
  Arms: 1
Drug: High Strength IDP-108 — Topical application once a day for 9 months
  Arms: 2
Drug: High Strength IDP-108 under occlusion — Topical application once a day for 9 months
  Arms: 3
Drug: Vehicle — Topical application once a day for 9 months
  Arms: 4

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of two concentrations of IDP-108 in treating patients with onychomycosis

ELIGIBILITY:
Inclusion Criteria:

* Presence of onychomycosis of the target toenail
* A positive fungal culture from the target toenail

Exclusion Criteria:

* Any disease or condition that might cause nail abnormalities or may interfere with clinical evaluations
* Presence of tinea pedis (athletes foot)
* Female subjects who are pregnant, nursing, planning a pregnancy, or become pregnant during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2007-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in area of infected nail | 9 months

SECONDARY OUTCOMES:
Change from baseline in mycological results | 9 months

CONTACTS AND LOCATIONS:
Locations (10):
- Mexico (10):
  - Unidad de Investigación en Salud, Chihuahua City, Chihuahua
  - Clinical Research Institute, Mexico City, Federal District
  - Hospital Central Militar, Mexico City, Federal District
  - Hospital General de México, México, Federal District
  - Instituto Dermatólogico de Jalisco "Dr. Jose Barba Rubio", Guadalajara, Jalisco
  - Hospital Dr. Ángel Leaño, Zapopan, Jalisco
  - MIRC/OCA Hospital, Monterrey, Nuevo León
  - Centro de Dermatología de Monterrey, Monterrey, Nuevo León
  - Hospital Universitario "José E. González", Monterrey, Nuevo León
  - Hospital Ignacio Morones Prieto SLP, San Luis Potosí City, San Luis Potosí

REFERENCES:
- [Derived] Tschen EH, Bucko AD, Oizumi N, Kawabata H, Olin JT, Pillai R. Efinaconazole solution in the treatment of toenail onychomycosis: a phase 2, multicenter, randomized, double-blind study. J Drugs Dermatol. 2013 Feb;12(2):186-92. PMID 23377392